CLINICAL TRIAL: NCT06535997
Title: Descriptive Cohort of French Patients Treated With Carbonetherapy Since October 2010 Outside PHRC-ETOILE - PRIMHADRON
Brief Title: Descriptive Cohort of French Patients Treated With Carbonetherapy Since October 2010 Outside PHRC-ETOILE
Acronym: PRIMHADRON
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Centre François Baclesse, Centre de lutte contre le cancer (CLCC) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0473
Record Dates: First submitted 2024-07-12; First posted 2024-08-02 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Cystic Carcinomas, Adenoid; Soft-tissue Sarcomas; Rhabdomyosarcoma Pleomorphic; Sarcoma,Soft Tissue; Osteosarcomas; Chondrosarcoma, Grade 3; Chordoma; Angiosarcomas
Keywords: Cancer; carbonetherapy; descriptive cohort
MeSH Terms: conditions — Neoplasms; Carcinoma, Adenoid Cystic; Sarcoma; Osteosarcoma; Chondrosarcoma; Lymphoma, Follicular; Chordoma; Hemangiosarcoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients traited for carbonetherapy outside the PHRC-ETOILE programme: Collection of clinical-biological data from medical records (retrospective). For patients alive, completion of a quality-of-life questionnaire and a medico-economic interview (prospective).
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — For patients alive only at the time of inclusion, completion of a quality-of-life questionnaire and a medico-economic interview (prospective).

SUMMARY:
Since the 1990s, carbonetherapy radiotherapy has been developed in a few sites around the world, mainly to treat inoperable and highly radioresistant tumors. In the absence of a treatment center of this type in France, the French health insurance system and health authorities (DGOS, INCa and HAS) have contributed to the setting up of a prospective randomized controlled study, PHRC-ETOILE, to evaluate this practice, and have also authorized, on the basis of expert opinion, treatment outside the PHRC of patients who could not be included in the PHRC but whose indications were very similar to those mentioned in the PHRC.

This "out-of-study" cohort began in October 2010, and has continued to grow steadily. By the end of 2022, it had reached 53 patients.

It is important to study the impact of carbonetherapy on these patients, in order to gain an initial appreciation of the benefits, tolerability and contribution of this practice for patients.

Local control, progression-free survival and overall survival in this cohort will be studied, as well as the role of carbon therapy in the management of these patients, some of whom are very complex. Complications attributable to carbon therapy, care pathways and changes in patients' quality of life will also be analyzed.

This analysis will make a contribution to the overall evaluation of carbonetherapy, assessing its usefulness and therefore the benefit to patients of its application. In our future prospects, some of these cases (around 23) could be used to consolidate the PHRC-ETOILE cohort.

This study will contribute to the development of the case for carbonetherapy, enabling the health authorities to make an informed decision on whether or not to expand access to this therapy.

* PHRC-ETOILE (First Transnational Randomized Prospective Trial Comparing Carbon Therapy versus Non-Carbon Therapy for Radioresistant Tumors)
* PHRC (Hospital clinical research programme)

ELIGIBILITY:
Inclusion Criteria :

* Patients aged ≥ 18 years at the time of inclusion
* Patients treated with Carbonetherapy outside PHRC-ETOILE from October 2010 to December 2023, after validation of their file by the health insurance expert, under an agreement providing for reimbursement for indications similar to those of PHRC-ETOILE for patients unable or unwilling to be included (re-irradiation, rare tumors or tumors of exceptional presentation not included in PHRC-ETOILE inclusion criteria). These include, by way of illustration :

  * Unresectable or non-operable cancers, or those with macroscopically incomplete resection (R2)
  * Radiation-resistant cancers considered eligible according to the following indicative list:
  * Cystic adenoid carcinomas (CAK) of the head and neck (excluding laryngeal and tracheal localizations)
  * Soft-tissue sarcomas
  * Pleiomorphic rhabdomyosarcomas only
  * Retroperitoneal sarcomas subject to technical feasibilitý - movement)
  * Osteosarcomas of any location and any grade
  * Chondrosarcomas (skull base excluded) grade greater than 2
  * Chordomas of the axial skeleton and pelvis (excluding skull base)
  * Angiosarcomas
* Patients who have not objected to the re-use of medical data for cancer research purposes, and who agree to be contacted by the investigator to complete the quality of life and care pathway questionnaires.

Exclusion Criteria:

* Refusal by the living patient to participate in research
* Failure to carry out initially planned carbon therapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients covered by the French Assurance Maladie from 2010 onwards for carbonetherapy treatment outside the PHRC-ETOILE programme
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Defined as the time elapsed between the start of carbonbased therapy and the date of the first event, i.e. 1st progression, 1st relapse or death (whatever the cause). Patients with no events by 12/31/2023 will be censored at the date of their last known tumor evaluation.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre François Baclesse, Centre de lutte contre le cancer (CLCC), Caen
  - Hôpital Michallon, CHU de Grenoble-Alpes, Grenoble

IPD SHARING:
Plan to Share IPD: Undecided
No final decision has been made yet regarding IPD sharing. The sponsor is currently reviewing institutional policies, data protection requirements and publication strategies. A plan may be implemented in the future depending on scientific interest and feasibility.